CLINICAL TRIAL: NCT01336660
Title: Phase 2/3 Study for Scorpion North Africa Middle East Envenomation With a Immune F(ab')2 (Equine) Antivenom Alacramyn NAMO. A Randomized, Double-Blind, Placebo-controlled, Prospective and Multicenter Study
Brief Title: A Trial of Equine F (ab')2 Antivenom for Treatment of Scorpion Envenomation in Morocco
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: Centre Antipoison et de Pharmacovigilane du Maroc (Unknown); Institut Pasteur du Maroc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XM-10/02
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Poisoning by Scorpion Sting
Keywords: Effectiveness; New Antivenom; North Africa and Middle East Scorpio Envenomation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine F(ab')2 antivenom (Experimental): Intensive care support and Equine F(ab')2 antivenom
  Interventions: Biological: Equine F(ab')2 antivenom
- Placebo (Placebo Comparator): Intensive care support plus placebo
  Interventions: Other: Intensive care support plus placebo

INTERVENTIONS:
Biological: Equine F(ab')2 antivenom — A single dose of 4 vials of Equine F(ab')2 antivenom will be administered intravenously over 10 minute
  Other Names: Alacramyn NA; Scorpion North Africa and Middle East Immune F(ab')2(Equine)
  Arms: Equine F(ab')2 antivenom
Other: Intensive care support plus placebo — Intensive care support as needed plus placebo
  Arms: Placebo

SUMMARY:
This study has the objective to demonstrate the effectiveness of Alacramyn NAMO in the treatment of North Africa and Middle East scorpions envenomation by reducing the severity of envenomation. The primary endpoint is make a comparison between antivenom and placebo groups, at 4 hours after study drug, of the number of cases showing improvement in class of envenomation.

DETAILED DESCRIPTION:
In an effort to shorten hospital stay and to further decrease mortality, a new antivenom has been developed. This antivenom is a third generation F(ab')2 "fabotherapeutic" agent.It is administered intravenously which should lead to rapid neutralization of circulating venom. This study will demonstrate whether or not use of the new antivenom in children receiving standardized supportive care leads to resolution of the syndrome within 4 hours of treatment.The onset of clinical symptoms following a scorpion envenomation is usually within 5 to 30 minutes following the sting.

Established a classification of the patient status to differentiate a simple scorpion sting from a severe envenomation. A simple sting (class I) is characterized by signs that are local only: pain at the inoculation point, redness, edema, and numbness.

A class II envenomation is characterized by the presence of some systemic signs: hypothermia, hyperthermia, chills, nausea, abdominal pain and diarrhea. Being 15 years old or younger or the presence of priapism, vomiting, sweating, or a body temperature greater than 39°C are factors predictive of severity.

A severe envenomation (class III) is characterized by cardiovascular failure, often leading to death; respiratory failure related to the cardiac failure; and neurologic failure due to hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 6 months to 15 years
* Class II B or III scorpion envenomation
* Presenting within 5 hours of sting
* Informed consent read and signed by parent or legal guardian

Exclusion Criteria:

* Unable to provide informed consent
* Prior use of antivenom for this envenomation
* Allergy to horse serum
* Pregnant or breast-feeding
* Patients with underlying condition mimicking symptoms of scorpion envenomation (congenital heart disease, chronic oxygen therapy, etcetera)

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2018-07-21 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
To demonstrate the effectiveness of Alacramyn NAMO in the treatment of scorpion envenomation by reducing the severity of envenomation | 4 hours after study drug
  Comparison between antivenom and placebo groups of the number of cases showing improvement in class of envenomation.

SECONDARY OUTCOMES:
Effectiveness of Alacramyn NAMO in the treatment of scorpion envenomation by reducing the severity of envenomation. | To 16 hours after treatment until discharge time and date
  Decrease in plasma venom levels from baseline to one hour after study drug administration; Respiratory rate (breaths per minute); Heart rate (beats per minute); Dose of dobutamine (cumulative, per hour);Incidence of cardiac failure; Incidence of ventilatory failure; Incidence of neurological failure; Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Walter Garcia, MD, Study Director — Instituto Bioclon; Rachida Soulaymani, Pr, Study Chair — Centre Antipoison et de Pharamacovigilance du Maroc; Sanae Achour, Principal Investigator — FES University Hospital; Asmae Khattabi, Study Chair — Ecole Nationale de Santé Publique
Locations (2):
- Morocco (2):
  - CHU Hassan II de Fès, Fes
  - Hôpital Ibn Zohr, Marrakech, Marrakesh

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided